CLINICAL TRIAL: NCT06825988
Title: The Use of the GRASP System for Postoperative Monitoring - a Feasibility Study
Brief Title: The Use of the GRASP System for Postoperative Monitoring
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other); Grasp AS (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 634183; Pilot Helse (Other Grant/Funding Number: Norwegian Research Council)
Record Dates: First submitted 2025-02-04; First posted 2025-02-13 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2023-11

CONDITIONS: Knee Arthroplasty, Total; Rehabilitation
Keywords: digital health; tangible interaction; postoperative monitoring; rehabilitation; knee arthroplasty; mixed methods; feasibility
MeSH Terms: interventions — Hand Strength

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Grasp system (Experimental): Grasp system (hardware and mobile application) during first 6 postsurgical weeks of rehabilitation. Subjects are instructed to report pain through squeezing the hardware in 3 different levels regulaly during the day, and, in addition enter answers to questions on patient reported outcome meassures (sleep quality, overall well-being, use of medication, appetit, physical activity) and register exercise time into the mobile application. Data entries will be presented as trajectories in graphs and charts in the app. At their 6 weeks physiotherapist consult, the physiotherapists will use the data during the consult.
  Interventions: Device: Grasp

INTERVENTIONS:
Device: Grasp — Grasp system (hardware and mobile application) during first 6 postsurgical weeks of rehabilitation. Subjects are instructed to report pain through squeezing the hardware in 3 different levels regulaly during the day, and, in addition enter answers to questions on patient reported outcome meassures (sleep quality, overall well-being, use of medication, appetit, physical activity) and register exercise time into the mobile application.

SUMMARY:
The aim of this study is to explore feasibility and user experience of a novel digital system containing a handheld electronic device and a mobile application - called Grasp - in the setting of postoperative monitoring of pain and patient reported outcome measures in knee arthroplasty patients.

The investigators will use a mixed-methods approach to gain in-depth insights into feasibility and user experience of this system in order to evaluate further improvement needs of both study design and intervention before a final randomised effect study. Feasibility will be evalutated through recruittment rates, adhererance to intervention protocol and study data sampling, and completion rates. Fidelity will be assessed as number of patients who are able to do as instructed in the protocol. In addition, the investigators will explore user experience through questionnaires after 2 and 6 weeks of use and through semi-structered interviews of participants and associated physiotherapists. Interviews will be transcribed for qualitative analyses.

ELIGIBILITY:
Inclusion Criteria:

* Elective joint arthroplasty
* Age: 30-70 years
* Must own and be able to use a smart phone
* Speak and understand Norwegian

Exclusion Criteria:

* Not able to give informed consent

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — gender definitions is not an exclusion criteria of this study.
Enrollment: 36 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of the intervention study | From enrollment to 6 weeks after surgery
  Feasibility of the intervention study will be evalutated through adhererance to intervention protocol. It will be assessed as number of patients who are able to do as instructed in the protocol. Fidilty >80% will be considered high, 50-80% moderate, and <50% low. The investigators expect a priori the adherance to protocol guidelines to decline during the 6 weeks intervention period
User experience | From enrollment to 6 weeks post surgery
  Mixed methods approach will be used to evaluate user experience. The investigators will make a mixed methods synthsis between participants questionnaires (by 2 and 6 weeks of intervention) and semi-structured interviews of up to 10 participants and associated physiotherapists by the end of the intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- Helse Bergen, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 2023-2038
Access Criteria: All documents are available on request